CLINICAL TRIAL: NCT03877926
Title: A Phase 3, Randomized, Double-blind, Parallel-group Trial to Evaluate the Lot Consistency, Immunogenicity, and Safety of AV7909 for Postexposure Prophylaxis of Anthrax in Healthy Adults
Brief Title: VELOCITY: An Anthrax Vaccine Clinical Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Emergent BioSolutions (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EBS.AVA.212
Record Dates: First submitted 2019-03-14; First posted 2019-03-18 (Actual); Results first posted 2021-12-21 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Anthrax
Keywords: Anthrax; AV7909; BioThrax; Bacillus anthracis; Anthrax Vaccine Adsorbed; Post-exposure Prophylaxis; Vaccine; CPG 7909; Adjuvant
MeSH Terms: conditions — Anthrax | interventions — Biothrax

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- AV7909 Lot 1 (Experimental): Participants meeting the entry criteria will be randomized 2:2:2:1 to one of four study groups. Groups 1 to 3 will each receive one of the three consecutively manufactured lots of AV7909, per the study visit schedule.
  Interventions: Biological: AV7909
- AV7909 Lot 2 (Experimental): Participants meeting the entry criteria will be randomized 2:2:2:1 to one of four study groups. Groups 1 to 3 will each receive one of the three consecutively manufactured lots of AV7909, per the study visit schedule.
  Interventions: Biological: AV7909
- AV7909 Lot 3 (Experimental): Participants meeting the entry criteria will be randomized 2:2:2:1 to one of four study groups. Groups 1 to 3 will each receive one of the three consecutively manufactured lots of AV7909, per the study visit schedule.
  Interventions: Biological: AV7909
- BioThrax (Active Comparator): Participants meeting the entry criteria will be randomized 2:2:2:1 to one of four study groups. In Group 4, one lot of BioThrax® vaccine will be administered, per the study visit schedule.
  Interventions: Biological: BioThrax

INTERVENTIONS:
Biological: AV7909 — AV7909 consists of Anthrax Vaccine Adsorbed (AVA) drug substance and CPG 7909 adjuvant. AVA drug substance in AV7909 is similar in composition and manufactured using the same process as commercial BioThrax® vaccine. BioThrax is licensed for post-exposure prophylaxis of anthrax disease. CPG 7909 is an immunostimulatory synthetic oligodeoxynucleotide that functions as an adjuvant. It is designed to induce an enhanced immune response.
  Arms: AV7909 Lot 1; AV7909 Lot 2; AV7909 Lot 3
Biological: BioThrax — BioThrax vaccine (Anthrax Vaccine Adsorbed; AVA) is licensed for post-exposure prophylaxis of anthrax disease.
  Arms: BioThrax

SUMMARY:
This study is designed to evaluate the lot consistency (using three consecutively manufactured lots), safety, and ability of the AV7909 anthrax vaccine to generate an immune response in healthy adults and compare the response to that induced by the currently licensed vaccine, BioThrax®, (Anthrax Vaccine Adsorbed; AVA) for post-exposure of anthrax disease.

DETAILED DESCRIPTION:
This is a Phase 3, multicenter, randomized, double-blind, parallel-group trial designed to evaluate the lot consistency (using three consecutively manufactured lots), immunogenicity, and safety of AV7909 administered in healthy adults for an indication of postexposure prophylaxis (PEP) of anthrax.

Healthy adults between 18 and 65 years of age (inclusive) will sign and date an informed consent form and then be screened for eligibility for participation in the study 2 to 28 days prior to randomization. Participants meeting the entry criteria will be randomized 2:2:2:1 to one of four study groups on Day 1. Randomization will be stratified by site.

Participants will be evaluated for safety through Day 64 [or the early withdrawal visit (EWV)], as assessed by clinical laboratory tests (hematology, serum chemistry, and urinalysis), monitoring of Adverse Events (AE) including Serious Adverse Events (SAE) and Adverse Events of Special Interest (AESI), vital signs, and physical examinations. Adverse Events of Special Interest are adverse events associated with autoimmune disease as defined by the Center for Biologics Evaluation and Research, and might represent a safety signal for vaccine-associated autoimmunity. Reactogenicity (solicited systemic and injection site reactions) will be assessed daily by the participants using electronic diaries (e-diaries) after each vaccination.

Information on the use of medications will be collected at each study visit. In addition, blood samples for auto-antibody assessment will be taken at Day 1 predose and Day 64 (or Early Withdrawal Visit).

Participants who receive at least one dose of vaccine but who for any reason discontinue vaccinations prematurely will be asked to participate in the further planned study visits up to Day 64 for safety assessment only.

Participants who receive at least one dose of vaccine will also be asked to participate in safety follow-up phone calls occurring on Day 43, Month 4, Month 7, Month 10, and Month 13 (nominally 0.5, 3, 6, 9, and 12 months after the last vaccination) to collect information on AEs, SAEs and any potential AESIs. Based on responses at these phone contacts, participants may be asked to return to the clinic for an unscheduled visit to provide blood samples for auto-antibody testing to investigate reports of potential AESIs.

Independent safety oversight will be provided by a Data Safety Monitoring Board, which will be notified of significant AEs as determined by the Medical Monitor on an ongoing basis.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained from the participant (dated and signed).
2. Healthy condition as established by medical history and clinical examination before entering into the study.
3. A male or female aged 18 to 65 years, inclusive, at the time of informed consent.
4. Body mass index (BMI) ≤35.0 kg/m^2 at Screening visit.
5. Have adequate venous access for phlebotomies.
6. For a woman of childbearing potential (WOCBP), negative serum pregnancy test at Screening and negative urine pregnancy test prevaccination on Day 1, not currently breastfeeding, and no intention to become pregnant during the study through Month 13. Every female participant is considered to be a WOCBP unless surgically sterile (bilateral oophorectomy or bilateral salpingectomy or hysterectomy) OR postmenopausal (defined as >12 consecutive months without menses and screening follicle-stimulating hormone >30 mIU/mL). Women who are not of childbearing potential are allowed to enroll if they are surgically sterile or postmenopausal as defined above.

Exclusion Criteria:

1. Use of any investigational or nonregistered product (drug, vaccine, device, or combination product) within 30 days preceding the dose of study vaccine, or planned use during the study through Month 13.
2. Positive test result on urine drug screen, any evidence of ongoing drug abuse or dependence (including alcohol), or recent history (over the past five years) of treatment for alcohol or drug abuse.
3. Chronic administration (defined as >14 days) of immunosuppressants or other immune-modifying drugs (includes oral or parenteral corticosteroids, for example, a glucocorticoid dose exceeding 10 mg/day prednisone or equivalent) within six months prior to the vaccine dose; inhalation use (for example, for seasonal allergies) is permitted.
4. Planned administration of any commercially-available vaccine from seven days prior to the first study vaccination through two weeks after the last vaccination.
5. Previous anaphylactic reaction, severe systemic response, or serious hypersensitivity to a prior immunization or a known allergy to synthetic Oligodeoxynucleotides, aluminum, formaldehyde, benzethonium chloride (phemerol), or latex.
6. History of anthrax disease, suspected exposure to anthrax, or previous vaccination with any anthrax vaccine.
7. Have a tattoo/scar/birthmark or any other skin condition affecting the deltoid area that may interfere with injection site assessments.
8. A positive blood test for hepatitis B surface antigen, hepatitis C antibody, or human immunodeficiency virus (HIV) HIV-1 or HIV-2 antibodies.
9. Any confirmed or suspected immunodeficiency condition (congenital or secondary) or autoimmune disease based on medical history and Physical Exam, for example, Guillain-Barré.
10. A family history of congenital or hereditary immunodeficiency.
11. Major congenital defects or serious chronic illness, including any cancer other than the following: a) any non-metastatic cancer (excluding hematologic malignancies) or melanoma of which the participant has been disease-free for at least five years and b) localized skin cancer, resected (including squamous cell and basal cell carcinomas).
12. Acute disease at the time of enrollment. Note that screening lab tests may be delayed to allow the resolution of a transient acute condition or the subject may be rescreened.
13. Any medical condition that, in the opinion of the investigator, could adversely impact the participant's participation or the conduct of the study.
14. Any planned elective surgery during the study through 12 months after the last vaccination.
15. Planned receipt of immunoglobulins and/or any blood products within the three months preceding study enrollment or at any point during the study period until after the final safety phone contact.
16. Woman of childbearing potential refusing to practice an adequate method of contraception from at least one month before Day 1 and continuing through Month 13.

    An adequate method of contraception is defined as abstinence from sexual intercourse; prior bilateral tubal ligation; monogamous relationship with a vasectomized partner (vasectomy performed at least six months prior to the participant's screening visit); or any of these forms of birth control: pill, intrauterine device (IUD), implantable or injectable contraceptive (for example, Norplant® or Depo-Provera®), removable device (for example, NuvaRing® or Evra® patch), or double-barrier method (condom with spermicide, diaphragm with spermicide). The Principal Investigator and/or designee will discuss with the participant the need to use adequate contraception consistently and correctly and document such conversation in the participant's chart. In addition, the Principal Investigator and/or designee will instruct the participant to call immediately if the selected contraception method is discontinued or if pregnancy is known or suspected.
17. Member or family member of the investigator site team.
18. Previously served in the military any time after 1990 and/or plan to enlist in the military at any time from screening through the final telephone contact.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3862 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2020-08-06 (Actual); Study Completion 2020-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gideon Akintunde, MD, Study Director — Emergent BioSolutions
Locations (35):
- United States (35):
  - Achieve Clinical Research, LLC, Birmingham, Alabama
  - Optimal Research, LLC, Huntsville, Alabama
  - Coastal Clinical Research, an AMR company, Mobile, Alabama
  - Central Phoenix Medical Clinic, LLC, Phoenix, Arizona
  - Clinical Research Consortium, an AMR company, Tempe, Arizona
  - California Research Foundation, San Diego, California
  - Optimal Research, LLC, San Diego, California
  - Research Centers of America, Hollywood, Florida
  - Optimal Research, LLC, Melbourne, Florida
  - New Horizon Research Center, Inc, Miami, Florida
  - Meridian Clinical Research, LLC, Savannah, Georgia
  - Advanced Clinical Research, Boise, Idaho
  - Christie Clinic, LLC, Champaign, Illinois
  - Optimal Research, LLC, Peoria, Illinois
  - The Iowa Clinic, PC, West Des Moines, Iowa
  - Heartland Research Associates, LLC, Augusta, Kansas
  - Hutchinson Clinic, Hutchinson, Kansas
  - Johnson County Clin-Trials, LLC, Lenexa, Kansas
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Benchmark Research New Orleans, Metairie, Louisiana
  - Optimal Research, LLC, Rockville, Maryland
  - The Center for Pharmaceutical Research, an AMR company, Kansas City, Missouri
  - Meridian Clinical Research, LLC, Omaha, Nebraska
  - Clinical Research Center of Nevada LLC, Las Vegas, Nevada
  - Rapid Medical Research, Inc., Cleveland, Ohio
  - Aventiv Research Inc., Grove City, Ohio
  - Lynn Institute of Norman, Norman, Oklahoma
  - Coastal Carolina Research Center, Inc, Mt. Pleasant, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Clinical Research Associates, Inc., Nashville, Tennessee
  - Tekton Research, Austin, Texas
  - Benchmark Research, Fort Worth, Texas
  - Benchmark Research San Angelo, San Angelo, Texas
  - Martin Diagnostic Clinic, Tomball, Texas
  - Advanced Clinical Research, West Jordan, Utah

REFERENCES:
- [Derived] Drobic B, Akintunde G, Kim J, Mirceta M, Beach M, Komlenovic V. Immunogenicity, safety, and lot consistency of the anthrax vaccine adsorbed, adjuvanted for post-exposure prophylaxis of anthrax in healthy adults: A phase 3, randomized, double-blind trial. Vaccine. 2026 Feb 6;72:128068. doi: 10.1016/j.vaccine.2025.128068. Epub 2025 Dec 15. PMID 41401704

RESULTS

PARTICIPANT FLOW:
Groups:
- AV7909 Lot 1: Eligible participants randomized to receive AV7909 Lot 1.
  AV7909: AV7909 consists of Anthrax Vaccine Adsorbed (AVA) drug substance and CPG 7909 adjuvant. AVA drug substance in AV7909 is similar in composition and manufactured using the same process as commercial BioThrax® vaccine. CPG 7909 is an immunostimulatory synthetic oligodeoxynucleotide that functions as an adjuvant.
- AV7909 Lot 2: Eligible participants randomized to receive AV7909 Lot 2.
  AV7909: AV7909 consists of Anthrax Vaccine Adsorbed (AVA) drug substance and CPG 7909 adjuvant. AVA drug substance in AV7909 is similar in composition and manufactured using the same process as commercial BioThrax vaccine. CPG 7909 is an immunostimulatory synthetic oligodeoxynucleotide that functions as an adjuvant.
- AV7909 Lot 3: Eligible participants randomized to receive AV7909 Lot 3.
  AV7909: AV7909 consists of Anthrax Vaccine Adsorbed (AVA) drug substance and CPG 7909 adjuvant. AVA drug substance in AV7909 is similar in composition and manufactured using the same process as commercial BioThrax vaccine. CPG 7909 is an immunostimulatory synthetic oligodeoxynucleotide that functions as an adjuvant.
- BioThrax: Eligible participants randomized to receive BioThrax vaccine.
  BioThrax vaccine (Anthrax Vaccine Adsorbed; AVA) is licensed for post-exposure prophylaxis of anthrax disease.
Period: Overall Study
Arm/Group | AV7909 Lot 1 | AV7909 Lot 2 | AV7909 Lot 3 | BioThrax
Started | 1103 | 1103 | 1098 | 558
Received at Least One Study Vaccination | 1100 | 1102 | 1097 | 558
Did Not Receive Any Study Vaccination | 3 | 1 | 1 | 0
Completed (Number of participants who completed 12-month follow-up after last study vaccination) | 1032 | 1026 | 1035 | 537
Not Completed | 71 | 77 | 63 | 21
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Death | 2 | 2 | 2 | 0
Not completed — Lost to Follow-up | 41 | 52 | 45 | 17
Not completed — Physician Decision | 2 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 18 | 21 | 12 | 4
Not completed — Other - Various | 4 | 1 | 1 | 0
Not completed — Not Treated | 3 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat Population (i.e., number of randomized participants) is used for baseline analysis.
Groups:
- AV7909 Lot 1: Eligible participants randomized to receive AV7909 Lot 1.
- AV7909 Lot 2: Eligible participants randomized to receive AV7909 Lot 2.
- AV7909 Lot 3: Eligible participants randomized to receive AV7909 Lot 3.
- BioThrax: Eligible participants randomized to receive BioThrax vaccine.
- Total: Total of all reporting groups
Arm/Group | AV7909 Lot 1 | AV7909 Lot 2 | AV7909 Lot 3 | BioThrax | Total
Number analyzed (Participants) | 1103 | 1103 | 1098 | 558 | 3862
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.0 (13.0) | 39.2 (13.1) | 38.9 (12.8) | 38.6 (12.4) | 39.0 (12.9)
Age, Customized [Count of Participants; unit: Participants]
  18-30 years | 341 | 355 | 352 | 176 | 1224
  31-50 years | 502 | 470 | 488 | 269 | 1729
  51-65 years | 260 | 278 | 258 | 113 | 909
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 650 | 615 | 647 | 308 | 2220
  Male | 453 | 488 | 451 | 250 | 1642
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race : American Indian or Alaska Native | 4 | 4 | 5 | 2 | 15
  Race : Asian | 17 | 18 | 24 | 15 | 74
  Race : Black or African American | 170 | 186 | 191 | 89 | 636
  Race : Native Hawaiian or Other Pacific Islander | 2 | 5 | 3 | 1 | 11
  Race : White | 878 | 865 | 852 | 439 | 3034
  Race : More than One Race | 22 | 20 | 14 | 9 | 65
  Race : Other | 8 | 3 | 5 | 1 | 17
  Race : Unknown | 2 | 2 | 4 | 2 | 10
  Ethnicity: Not Hispanic or Latino | 910 | 938 | 945 | 450 | 3243
  Ethnicity: Hispanic or Latino | 177 | 156 | 142 | 98 | 573
  Ethnicity: Unknown | 4 | 2 | 8 | 4 | 18
  Ethnicity: Not Reported | 12 | 7 | 3 | 6 | 28
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1103 | 1103 | 1098 | 558 | 3862
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.9 (4.3) | 27.3 (4.3) | 27.2 (4.3) | 27.3 (4.2) | 27.1 (4.3)

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titer (GMT) of Toxin Neutralizing Antibody (TNA) 50% Neutralization Factor (NF50) at Day 64
Description: GMT of TNA NF50 at Day 64 in AV7909 study groups (Lots 1, 2 and 3) and BioThrax group. The outcome measure in AV7909 study groups was assessed for AV7909 lot-to-lot consistency, which was based on GMT TNA NF50 response at Day 64, wherein the 95% confidence interval (CI) for ratios of geometric mean titer (GMT) of TNA NF50 at Day 64 (seven weeks after second AV7909 vaccination) for each of the three AV7909 lot-to-lot comparisons had to be within equivalence margin of 0.5 and 2.0.
Time Frame: Day 64 (seven weeks after second AV7909 vaccination)
Population: Participants that met protocol-defined immunogenicity criteria from AV7909 Lot 1 group (n=878), AV7909 Lot 2 group (n=896), AV7909 Lot 3 group (n=896) and BioThrax group (n=454) are included.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer (TNA NF50)
Groups:
- AV7909 Lot 1: Eligible participants who received AV7909 vaccine lot 1.
- AV7909 Lot 2: Eligible participants who received AV7909 vaccine lot 2.
- AV7909 Lot 3: Eligible participants who received AV7909 vaccine lot 3.
- BioThrax: Eligible participants who received BioThrax vaccine.
Arm/Group | AV7909 Lot 1 | AV7909 Lot 2 | AV7909 Lot 3 | BioThrax
Number analyzed (Participants) | 878 | 896 | 896 | 454
Titer (TNA NF50) | 0.753 [0.708 to 0.800] | 0.746 [0.703 to 0.791] | 0.718 [0.676 to 0.763] | 0.335 [0.305 to 0.368]
Statistical Analysis 1: Comparison: AV7909 Lot 1 vs AV7909 Lot 2; Test type: Equivalence — The 95% CIs for the Day 64 TNA NF50 GMT ratios between AV7909 Lot 1 and Lot 2 had to be within 0.5 to 2.0 equivalence margin; Ratio = 1.01, 95% CI 2-sided [0.93 to 1.10]
Statistical Analysis 2: Comparison: AV7909 Lot 1 vs AV7909 Lot 3; Test type: Equivalence — The 95% CIs for the Day 64 TNA NF50 GMT ratios between AV7909 Lot 1 and Lot 3 had to be within 0.5 to 2.0 equivalence margin; Ratio = 1.05, 95% CI 2-sided [0.96 to 1.14]
Statistical Analysis 3: Comparison: AV7909 Lot 2 vs AV7909 Lot 3; Test type: Equivalence — The 95% CIs for the Day 64 TNA NF50 GMT ratios between AV7909 Lot 2 and Lot 3 had to be within 0.5 to 2.0 equivalence margin; Ratio = 1.04, 95% CI 2-sided [0.95 to 1.13]

2. Primary Outcome: Percentage of Participants in AV7909 Lot 1, Lot 2 and Lot 3 Groups Achieving a TNA NF50 ≥0.56 on Day 64
Description: Proportion of participants with TNA NF50 ≥0.56 at Day 64 in each AV7909 study groups (Lot 1, Lot 2, Lot 3). The assessment of the immune response in each study group was pre-defined as the lower bound of the two-sided 95% CI to be ≥40% for the percentage of AV7909 participants in each of the three lots achieving a TNA NF50 ≥0.56 at seven weeks after second AV7909 vaccination (Day 64).
Time Frame: Day 64 (seven weeks after second AV7909 vaccination)
Population: Data from participants that met protocol-defined criteria for inclusion in the immunogenicity population are included in the analysis; i.e., AV7909 Lot 1 n=878; AV7909 Lot 2 n=896; AV7909 Lot 3 n=896. Pre-defined success criteria (lower bound of the two-sided 95% CI to be ≥40% for the percentage of participants achieving a TNA NF50 ≥0.56 at Day 64) was only applicable for AV7909 study groups and not for BioThrax group; therefore, BioThrax group is not included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AV7909 Lot 1 | AV7909 Lot 2 | AV7909 Lot 3
Number analyzed (Participants) | 878 | 896 | 896
percentage of participants | 68.5 [65.3 to 71.5] | 66.1 [62.9 to 69.2] | 64.5 [61.3 to 67.6]

3. Primary Outcome: Percentage of AV7909 Participants Achieving a TNA NF50 ≥0.56 on Day 64
Description: Percentage of AV7909 participants (from all three AV7909 study groups pooled) achieving a TNA NF50 ≥0.56 on Day 64 (seven weeks after second AV7909 vaccination). The assessment of the immune response in AV7909 participants was pre-defined as the lower bound of the two-sided 95% CI for proportion of AV7909 participants with TNA NF50 ≥0.56 at Day 64 ≥40%.
Time Frame: Day 64 (seven weeks after second AV7909 vaccination)
Population: Data from participants who met protocol-defined criteria for inclusion in the immunogenicity population from all three AV7909 study groups (i.e., pooled AV7909; n=2670) were used for the analysis. The pre-defined success criteria (lower bound of the two-sided 95% CI to be ≥40% for the percentage of participants achieving a TNA NF50 ≥0.56 on Day 64) was not applicable for BioThrax participants, therefore BioThrax group was not included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Pooled AV7909: Participants from groups 1-3 [.e., AV7909 Lot 1 (group 1), AV7909 Lot 2 (group 2) and AV7909 Lot 3 (group 3)] were pooled to assess TNA NF50 response at Day 64.
Arm/Group | Pooled AV7909
Number analyzed (Participants) | 2670
percentage of participants | 66.3 [64.5 to 68.1]
Statistical Analysis 1: Comparison: Pooled AV7909; Test type: Other; Percentage of participants = 66.3, 95% CI 2-sided [64.5 to 68.1]

4. Primary Outcome: Percentage of AV7909 Participants and BioThrax Participants With TNA NF50 ≥0.29 at Day 64
Description: Proportion of AV7909 participants (in each AV7909 study groups) and BioThrax participants who achieved TNA NF50 ≥0.29 at Day 64. Non-inferiority of AV7909 vaccine to BioThrax vaccine at Day 64 was assessed as determined by the two-sided lower bound for the 95% CI of the difference in the percentage of AV7909 participants (three lots pooled) with a TNA NF50 ≥0.29 and the percentage of BioThrax participants with a TNA NF50 ≥0.29 being greater than -15%.
Time Frame: Day 64 (seven weeks after second AV7909 vaccination; five weeks after third BioThrax vaccination)
Population: Data from participants who met protocol-defined criteria for inclusion in the immunogenicity population from each AV7909 study group (Lot 1 n=878; Lot 2 n=896; Lot 3 n=896) and BioThrax group (n=454) were used in the analysis. For the non-inferiority assessment, participants who met pre-defined criteria (achievement of TNA NF50 ≥0.29 at Day 64) from the pooled AV7909 study groups 1-3 (AV7909 Lot 1, Lot 2, Lot 3; i.e., Pooled AV7909) and BioThrax group were included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- AV7909 Lot 1: Eligible participants who received AV7909 vaccine lot 1 and achieved TNA NF50 ≥0.29 at Day 64.
- AV7909 Lot 2: Eligible participants who received AV7909 vaccine lot 2 and achieved TNA NF50 ≥0.29 at Day 64.
- AV7909 Lot 3: Eligible participants who received AV7909 vaccine lot 3 and achieved TNA NF50 ≥0.29 at Day 64.
- BioThrax: Eligible participants who received BioThrax vaccine and achieved TNA NF50 ≥0.29 at Day 64.
Arm/Group | AV7909 Lot 1 | AV7909 Lot 2 | AV7909 Lot 3 | BioThrax
Number analyzed (Participants) | 878 | 896 | 896 | 454
percentage of participants | 86.9 [84.5 to 89.1] | 87.2 [84.8 to 89.3] | 85.8 [83.4 to 88.0] | 62.1 [57.5 to 66.6]
Statistical Analysis 1: Comparison: AV7909 Lot 1 vs AV7909 Lot 2 vs AV7909 Lot 3 vs BioThrax; Test type: Non-Inferiority — A non-inferiority margin of -15% was used for the difference in percentage of AV7909 participants (pooled from three AV7909 study groups [Lot 1, 2, and 3]) vs. BioThrax participants who achieved TNA NF50 ≥0.29 at Day 64. The success criterion was defined as the lower bound of 95% confidence interval of the difference in the percentage of AV7909 vs. BioThrax participants being greater than -15%; Difference in percentage = 24.5, 95% CI 2-sided [20.0 to 29.2]

5. Primary Outcome: Incidence of Serious Adverse Events
Description: Number of AV7909 participants or BioThrax participants who received at least one vaccination and reported serious adverse event(s) (SAEs) from the time of the first vaccination on Day 1 through Day 394.
Time Frame: Day 1 though Day 394
Population: For the relative risk of SAE incidence analysis, participants from all three AV7909 study groups (Lot 1, Lot 2, Lot 3) since AV7909 lots 1, 2 and 3 were considered the same product (consecutively manufactured, and released with the same product specifications); hence, it was pre-defined to combine SAE data from participants across the three AV7909 lots for SAE relative risk analysis.
Measure: Count of Participants; unit: Participants
Groups:
- AV7909 Lot 1: Eligible participants who received at least one dose of AV7909 Lot 1.
- AV7909 Lot 2: Eligible participants who received at least one dose of AV7909 Lot 2.
- AV7909 Lot 3: Eligible participants who received at least one dose of AV7909 Lot 3.
- BioThrax: Eligible participants who received at least one dose of BioThrax vaccine.
Arm/Group | AV7909 Lot 1 | AV7909 Lot 2 | AV7909 Lot 3 | BioThrax
Number analyzed (Participants) | 1100 | 1102 | 1097 | 558
Participants | 21 | 16 | 21 | 4
Statistical Analysis 1: Comparison: AV7909 Lot 1 vs AV7909 Lot 2 vs AV7909 Lot 3 vs BioThrax; Test type: Other — Relative risk of serious adverse events incidence between AV7909 (combined from all three AV7909 lots) and BioThrax; Relative risk (AV7909/BioThrax) = 2.5, 95% CI 2-sided [0.9 to 6.5] — The 95% CI of the relative risk was derived using the Farrington-Manning relative risk score statistic

6. Secondary Outcome: Percentage of AV7909 Participants Achieving a TNA NF50 ≥0.15 on Day 29.
Description: Proportion of AV7909 participants (in each AV7909 study group) who achieved TNA NF50 ≥0.15 at Day 29 (two weeks after second AV7909 vaccination). Assessment of the lower bound of the two-sided 95% CI to be ≥67% for the percentage of AV7909 participants in AV7909 study groups 1-3 (Pooled AV7909) achieving a TNA NF50 ≥0.15 on Day 29 was performed.
Time Frame: Day 29 (two weeks after second AV7909 vaccination)
Population: Data from participants who met protocol-defined criteria for inclusion in the immunogenicity population (AV7909 study groups 1-3) were used in the analysis. The pre-defined success criteria (lower bound of the two-sided 95% CI to be ≥67% for the percentage of participants achieving a TNA NF50 ≥0.15 on Day 29) was not applicable for BioThrax, therefore BioThrax group was not included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- AV7909 Lot 1: Eligible participants who received AV7909 vaccine lot 1 and achieved TNA NF50 ≥0.15 at Day 29.
- AV7909 Lot 2: Eligible participants who received AV7909 vaccine lot 2 and achieved TNA NF50 ≥0.15 at Day 29.
- AV7909 Lot 3: Eligible participants who received AV7909 vaccine lot 3 and achieved TNA NF50 ≥0.15 at Day 29.
Arm/Group | AV7909 Lot 1 | AV7909 Lot 2 | AV7909 Lot 3
Number analyzed (Participants) | 863 | 878 | 876
percentage of participants | 98.1 [97.0 to 98.9] | 97.9 [96.8 to 98.8] | 97.4 [96.1 to 98.3]
Statistical Analysis 1: Comparison: AV7909 Lot 1 vs AV7909 Lot 2 vs AV7909 Lot 3; Test type: Other — Success criteria was defined as the lower bound for the 95% CI for the proportion of participants pooled from all three AV7909 study groups with TNA NF50 ≥0.15 to be ≥67%; Percentage of participants = 97.8, 95% CI 2-sided [97.2 to 98.3]

7. Secondary Outcome: Incidence of Adverse Events
Description: Number of AV7909 or BioThrax participants who received at least one vaccination and had at least one adverse event reported from the time of the first vaccination on Day 1 through Day 64.
Time Frame: Day 1 through Day 64
Population: Data from participants who received at least one dose of AV7909 vaccine Lot 1 (n=1100), Lot 2 (n=1102) or Lot 3 (n=1097) or BioThrax vaccine (n=558) are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | AV7909 Lot 1 | AV7909 Lot 2 | AV7909 Lot 3 | BioThrax
Number analyzed (Participants) | 1100 | 1102 | 1097 | 558
Participants | 410 | 400 | 408 | 210

8. Secondary Outcome: Incidence of Adverse Events of Special Interest (Events of Autoimmune Etiology)
Description: Incidence of adverse events of special interest (AESIs; events of autoimmune etiology) from the time of the first vaccination on Day 1 through Day 394 in participants who received at least one dose of AV7909 (Lot 1, Lot 2 or Lot 3) or BioThrax vaccines.
Time Frame: Day 1 through Day 394
Population: Data from participants who received at least one dose of AV7909 vaccine (Lot 1, Lot 2 or Lot 3) or BioThrax vaccine are used in the analysis. Since AV7909 lots 1, 2 and 3 were considered the same product (consecutively manufactured, and released with the same product specifications), it was pre-defined to combine AESI data from participants across the three AV7909 lots for AESI relative risk analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | AV7909 Lot 1 | AV7909 Lot 2 | AV7909 Lot 3 | BioThrax
Number analyzed (Participants) | 1100 | 1102 | 1097 | 558
Participants | 5 | 4 | 6 | 2
Statistical Analysis 1: Comparison: AV7909 Lot 1 vs AV7909 Lot 2 vs AV7909 Lot 3 vs BioThrax; Test type: Other — Relative risk of adverse events of special interest (events of autoimmune etiology) incidence between AV7909 (combined from all three AV7909 lots) and BioThrax; Relative risk (AV7909/BioThrax) = 1.3, 95% CI 2-sided [0.3 to 5.0] — The 95% CI of the relative risk was derived using the Farrington-Manning relative risk score statistic

9. Secondary Outcome: Incidence of Solicited Systemic Reactogenicity Events
Description: Incidence of any solicited systemic reactogenicity reaction after any AV7909 or BioThrax vaccination.
Time Frame: Day 1-7, Day 15-21, Day 29-35 (within 7 days after each vaccination, inclusive of the vaccination day)
Population: Data from participants (solicited systemic reactogenicity events after any vaccination) who received at least one dose of AV7909 vaccine or BioThrax vaccine are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | AV7909 Lot 1 | AV7909 Lot 2 | AV7909 Lot 3 | BioThrax
Number analyzed (Participants) | 1100 | 1102 | 1097 | 558
Participants | 930 | 923 | 906 | 438

10. Secondary Outcome: Incidences of Solicited Injection Site Reactogenicity Events
Description: Incidence of any solicited injection site reactogenicity reaction after any AV7909 (Lots 1, 2 or 3) or BioThrax vaccination.
Time Frame: Day 1-7, Day 15-21, Day 29-35 (within 7 days after each vaccination, inclusive of the vaccination day)
Population: Data from participants who received at least one dose of AV7909 or BioThrax dose are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | AV7909 Lot 1 | AV7909 Lot 2 | AV7909 Lot 3 | BioThrax
Number analyzed (Participants) | 1100 | 1102 | 1097 | 558
Participants | 1009 | 1010 | 1013 | 525

ADVERSE EVENTS:
Time Frame: Day 1 through Day 394.
Description: Adverse events, serious adverse events and adverse events of special interest (events of autoimmune etiology) were collected from Day 1 through Day 394. Local and systemic reactogenicity were solicited for seven days after each vaccination.
Arm/Group | AV7909 Lot 1 | AV7909 Lot 2 | AV7909 Lot 3 | BioThrax
All-Cause Mortality (participants affected / at risk) | 2/1100 | 2/1102 | 2/1097 | 0/558
Serious Adverse Events (participants affected / at risk) | 21/1100 | 16/1102 | 21/1097 | 4/558
Other Adverse Events (participants affected / at risk) | 193/1100 | 189/1102 | 120/1097 | 110/558
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AV7909 Lot 1 (N=1100) | AV7909 Lot 2 (N=1102) | AV7909 Lot 3 (N=1097) | BioThrax (N=558)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal prolapse (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Treatment noncompliance (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Corona virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vulval abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sialoadenitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 2 (2) | 0 (0) | 1 (1)
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphemia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular disorders (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AV7909 Lot 1 (N=1100) | AV7909 Lot 2 (N=1102) | AV7909 Lot 3 (N=1097) | BioThrax (N=558)
Diarrhoea (Gastrointestinal disorders) | 10 (10) | 5 (6) | 7 (8) | 6 (6)
Injection site pain (General disorders) | 32 (57) | 35 (57) | 29 (54) | 13 (32)
Injection site erythema (General disorders) | 5 (6) | 8 (8) | 16 (16) | 9 (9)
Injection site induration (General disorders) | 10 (11) | 11 (11) | 8 (9) | 54 (69)
Injection site swelling (General disorders) | 5 (6) | 5 (5) | 8 (9) | 15 (16)
Injection site warmth (General disorders) | 5 (6) | 2 (3) | 5 (5) | 7 (8)
Injection site bruising (General disorders) | 5 (6) | 5 (5) | 1 (1) | 9 (10)
Injection site pruritus (General disorders) | 4 (5) | 2 (3) | 3 (3) | 13 (14)
Injection site mass (General disorders) | 1 (1) | 2 (2) | 0 (0) | 8 (10)
Upper respiratory tract infection (Infections and infestations) | 27 (30) | 34 (36) | 31 (34) | 12 (14)
Urinary tract infection (Infections and infestations) | 18 (21) | 13 (18) | 21 (23) | 4 (4)
Nasopharyngitis (Infections and infestations) | 12 (12) | 8 (8) | 10 (10) | 6 (7)
Influenza (Infections and infestations) | 8 (8) | 6 (6) | 7 (7) | 6 (6)
Vaccination complication (Injury, poisoning and procedural complications) | 27 (29) | 31 (33) | 28 (31) | 7 (8)
Procedural headache (Injury, poisoning and procedural complications) | 20 (21) | 26 (27) | 31 (34) | 12 (14)
Musculoskeletal procedural complication (Injury, poisoning and procedural complications) | 14 (14) | 21 (21) | 26 (28) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 18 (20) | 10 (10) | 9 (9) | 6 (6)
Headache (Nervous system disorders) | 16 (17) | 15 (17) | 14 (15) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2019-03-14): https://cdn.clinicaltrials.gov/large-docs/26/NCT03877926/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-15): https://cdn.clinicaltrials.gov/large-docs/26/NCT03877926/SAP_001.pdf
  • Informed Consent Form (2019-01-29): https://cdn.clinicaltrials.gov/large-docs/26/NCT03877926/ICF_003.pdf